CLINICAL TRIAL: NCT00466375
Title: Genetic Basis of Hemangiomas
Status: Terminated | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Beth A Drolet, MD, Professor and Vice Chairman of Pediatric Dermatology, Medical College of Wisconsin
Other Study IDs: Genetics of Hemangioma
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Hemangioma, Vascular Anomalies
Keywords: hemangioma; vascular anomaly; infantile hemangioma
MeSH Terms: conditions — Hemangioma; Vascular Malformations; Hemangioma, Capillary | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Buccal smear (cheek cells)or small blood sample (4 mL or one teaspoon)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Patients with a hemangioma.
  Interventions: Genetic: Cheek cell samples or blood sample (4mL)
- B.: Patients with a vascular anomaly.
  Interventions: Genetic: Cheek cell sample or blood sample (4mL)

INTERVENTIONS:
Genetic: Cheek cell samples or blood sample (4mL) — DNA will be extracted from cheek cell or blood samples from parents and child having hemangioma.
  Groups: A
Genetic: Cheek cell sample or blood sample (4mL) — DNA will be extracted from cheek cell or blood samples of parents and child with a vascular anomaly.
  Groups: B.

SUMMARY:
The purpose of this study is to determine if there are genes that are common in children with infantile hemangioma. This information will allow physicians to improve care for patients who have been diagnosed with this disease and to provide their parents with more complete information regarding the cause of this disease. This research is being done because many unanswered questions remain regarding children with infantile hemangioma. There are very few medications to treat infants with hemangiomas.

DETAILED DESCRIPTION:
WHAT IS INVOLVED IN THE RESEARCH STUDY?

* Buccal smear (cheek cells) or small blood sample (4 mL or 1 teaspoon) from child being seen in the Dermatology clinic having infantile hemangioma or vascular anomaly
* Buccal smear (cheek cells) or small blood sample (4 mL or 1 teaspoon) from parents of child

If you and your child agree to be in this study, the following will happen:

1. Informed consent and permission to use or disclose your/your child's health information for research purposes will be obtained by Dr. Drolet, the principal investigator, or her research team. You will receive a copy of this consent form.
2. A buccal swab or blood sample will be obtained from you and your child; buccal sampling involves rubbing the inside of your cheek and removing cells to perform a genetic test called "Genomewide Association (GWA).

We expect you and your child to be involved in this study until you and your child have the genetic testing performed.

ELIGIBILITY:
Study Population Inclusion Criteria:

* No limit to age
* Diagnosis of infantile hemangioma and/or vascular anomaly
* Unaffected twin sibling
* Each patient's authorized legal guardian must understand the nature of the study and must provide written informed consent. Each patient must also give assent to study participation.

Study Population Exclusion Criteria:

* Diagnosis other than infantile hemangioma or vascular anomaly
* If the lesion has resolved and cannot be confirmed as a hemangioma by clinical exam
* If the biologic parents are unwilling or unable to submit DNA samples the child will be excluded from the DNA study. Therefore, if DNA samples cannot be or are not obtained from both biologic parents, the child and family will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinics from Children's Hospital of Wisconsin.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2007-04; Primary Completion 2014-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
SNP | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Beth Drolet, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States